CLINICAL TRIAL: NCT04239144
Title: Role of Sympathetic Denervation by Video-assisted Thoracoscopy in Control of Cardiac Arrhythmias in Patients With Chagas Disease - Pilot Study Randomized Controlled Trial
Brief Title: Sympathetic Denervation by Video-assisted Thoracoscopy in Control of Cardiac Arrhythmias in Patients With Chagas Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Paulo Manuel Pêgo Fernandes, Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49701215.2.0000.0068
Record Dates: First submitted 2019-01-23; First posted 2020-01-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chagas Cardiomyopathy; Ventricular Arrythmia
Keywords: Ventricular Tachycardia,; Chagas Disease; Catheter Ablation; Bilateral Sympathectomy; Cardiac Sympathetic Denervation
MeSH Terms: conditions — Chagas Cardiomyopathy; Tachycardia, Ventricular; Chagas Disease | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: In this pilot study, the investigators will select 45 patients with Chagas cardiomyopathy with ICD who presented at least four ICD therapies in the prior six months. These patients will be randomly assigned to three groups, 15 patients in medical therapy group, 15 in catheter ablation and 15 in bilateral sympathectomy. The objective of this study is to evaluate the efficacy of the bilateral sympathectomy in the reduction of ventricular tachycardia in patients with Chagas cardiomyopathy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical therapy group (No Intervention): Arm 1 - 15 patients allocated to this group will receive conventional antiarrhythmic medical treatment according the guidelines with additional impregnation of amiodarone, incremental dose of beta-blocker and if possible ICD reprograming.
- Catheter ablation (Active Comparator): Intervention Arm 2 -15 patients allocated to this group will undergo epicardial and endocardial catheter ablation with the use of irrigated contact sensor tip catheter. Voltage electroanatomical mapping using Carto System will be performed in all cases and if hemodynamically stable VT is induced, activation mapping will also be performed. The result of ablation will be defined as (1) complete success (all VTs non-inducible); (2) partial success (clinical VT non inducible, but other morphologies still inducible) and (3) failure (clinical VT still inducible).
  Interventions: Procedure: Catheter ablation
- Bilateral sympathectomy (Experimental): Interventional Arm 3 - 15 patients allocated to this group will undergo bilateral sympathectomy, which will be performed using video assisted thoracoscopy using the Ethicon Ultracision device. The denervation consists of lower 1/3 stellate ganglion and T3- T4 thoracic interspinal space videothoracoscopic cutting, isolating the whole sympathetic chain between these two points using ultracision device on the nerve branches. The cephalic portion of the stellate ganglion will be preserved to avoid Horner's syndrome and the electrocautery use will also be avoided for the same reason. Hemodynamic and echocardiographic behaviors will be continuously monitored during these surgical maneuvers.
  Interventions: Procedure: Bilateral sympathectomy

INTERVENTIONS:
Procedure: Bilateral sympathectomy — Bilateral sympathectomy will be performed using video assisted thoracoscopy using the Ethicon Ultracision device. The denervation consisted of left lower 1/3 stellate ganglion and T3- T4 thoracic interspinal space videothoracoscopic cutting, isolating the whole sympathetic chain between these two points using ultracision device on the nerve branches. The cephalic portion of the stellate ganglion was preserved to avoid Horner's syndrome and the electrocautery use was also avoided due to the same reason. The nerve was blocked using Ultracision device to avoid thermic lesion of the stellate ganglion. Hemodynamic and echocardiographic behaviors were continuously monitored during these surgical maneuvers.
  Other Names: Cardiac Sympathetic Denervation
  Arms: Bilateral sympathectomy
Procedure: Catheter ablation — Catheter ablation - patients allocated to this group will undergone epicardial and endocardial catheter ablation with the use of irrigated contact sensor tip catheter. Voltage electroanatomical mapping using Carto System will be performed in all cases and if hemodynamically stable VT is induced activation mapping will also be performed. The aim of the ablation is to eliminate the clinical VT additionally to substrate modification. The result of ablation will be defined as (1) complete success; (2) partial success and (3) failure.
  Arms: Catheter ablation

SUMMARY:
Ventricular tachycardia (VT) is the main cause of sudden death in patients with structural heart diseases. The use of ICD (implantable cardio-defibrillator) could prevent sudden death, however, the occurrence of repetitive shock decreases significantly the quality of life and could increase the mortality rate. Chagas disease in our environment is the most common heart disease and often associated with the occurrence appropriate ICD therapies.

The chronic treatment of VT aims to prevent recurrences with the use of antiarrhythmic drugs and catheter ablation, but in many cases, these treatments are insufficient to control the VT. Cardiac Sympathetic Denervation by bilateral sympathectomy has been described as an alternative treatment of VT refractory to medical treatment and radiofrequency ablation, especially in patients with channelopathies. This treatment could have a role in patients with structural heart disease.

The objective of this study is to evaluate the efficacy of the bilateral sympathectomy in the reduction of ventricular tachycardia in patients with Chagas cardiomyopathy. In this pilot study, the investigators will select 45 patients with Chagas cardiomyopathy with ICD who presented at least four ICD therapies in the prior six months. These patients will be randomly assigned to three groups, 15 patients in medical therapy group, 15 in catheter ablation and 15 in bilateral sympathectomy.

DETAILED DESCRIPTION:
OBJECTIVE

Primary

• Evaluate the efficacy of bilateral sympathectomy in the reduction of VT episodes in patients with Chagas cardiomyopathy.

Secondary

* To compare the efficacy of bilateral sympathectomy against VT ablation and against optimal medical therapy.
* To evaluate the density of ventricular premature beats 24-hour Holter and monitor the events recorded by the ICD and the impact of the treatment performed.
* To evaluate the length of the hospital stay according to the type of intervention.
* To evaluate the rate of clinical complications according to the type of intervention.
* To evaluate the impact of treatment on left ventricular function.

Follow up

Outcomes Assessment in six months and one year

* Recurrence rate of appropriate therapies;
* Density of ventricular ectopies;
* Complication rates per type of intervention;
* Number of in-hospital days per type of intervention;
* Assessment of LV function;

METHODS

This is a pilot, single-centre, open-label, randomized trial in patients with Chagas disease and multiple appropriate ICD therapies. This study consists of three groups: (1) medical treatment, (2) catheter ablation and (3) bilateral sympathectomy, being included 15 patients in each group.

Inclusion Criteria:

* Patients with Chagas Disease Cardiomyopathy having an ICD
* At least four appropriate ICD therapies in the past six months, documented by device interrogation or medical records;
* Use of amiodarone and beta blockers in an optimized fashion;
* Life expectancy of more than one year
* Conditions for following the plan of clinical follow-up of the study.

Exclusion criteria:

* Presence of an absolute contraindication to receive any of the possible treatments of the study;
* Pregnant Woman;
* Less than 18 years-old;
* Renal insufficiency with creatinine >2.5 mg/dL (221 umol/L);
* Mobile thrombus in the left ventricle;
* Left Ventricle Ejection fraction < 10%;
* Unstable angina;
* Severe aortic stenosis
* Primary severe mitral insufficiency;
* New York Heart Association (NYHA) functional class IV;
* Previous cardiac surgery or scheduled.

The patients will be recruited consecutively in the outpatient clinic of Cardiac Pacing Unit, or in outpatient clinic of Arrhythmias Clinical Unit or in the Emergency Clinical Unit.

Group 1 - Medical Treatment: patients allocated to this group will receive amiodarone reimpregnation, incremental dose of beta-blocker and if possible ICD reprogramming.

Group 2 - Catheter ablation: patients allocated to this group will undergo epicardial and endocardial catheter ablation with the use of an irrigated contact sensor tip catheter. Voltage electroanatomical mapping using Carto System will be performed in all cases and if hemodynamically stable VT is induced, activation mapping will also be performed. The aim of the ablation is to eliminate the clinical VT additionally to substrate modification. The result of ablation will be defined as (1) complete success (all VTs non-inducible); (2) partial success (clinical VT non inducible, but other morphologies still inducible) and (3) failure (clinical VT still inducible).

Group 3 - Bilateral sympathectomy - bilateral sympathectomy will be performed using video assisted thoracoscopy using the Ethicon Ultracision device. The denervation consists of lower 1/3 stellate ganglion and T3- T4 thoracic interspinal space videothoracoscopic cutting, isolating the whole sympathetic chain between these two points using ultracision device on the nerve branches. The cephalic portion of the stellate ganglion will be preserved to avoid Horner's syndrome and the electrocautery use will also be avoided for the same reason. Hemodynamic and echocardiographic behaviors will be continuously monitored during these surgical maneuvers. After the application, 10 ml of 0.25% bupivacaine solution will be injected along the site of the pleural dissection for postoperative analgesia. The lung will be reinflated under direct vision and a small tube will be inserted to remove the air through the upper incision, which will be removed at the end of the operation if possible. The two port sites will be closed primarily with absorbable stitches.

The study conformed to the principles outlined in the Declaration of Helsinki and was approved by the ethics committee and institutional review board of our hospital. All patients will provide written informed consent before randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chagas Disease Cardiomyopathy having an ICD
* At least four appropriate ICD therapies in the past six months, documented by device interrogation or medical records;
* Use of amiodarone and beta blockers in an optimized fashion;
* Life expectancy of more than one year
* Conditions for following the plan of clinical follow-up of the study.

Exclusion criteria:

* Presence of an absolute contraindication to receive any of the possible treatments of the study;
* Pregnant Woman;
* Less than 18 years-old;
* Renal insufficiency with creatinine >2.5 mg/dL (221 umol/L);
* Mobile thrombus in the left ventricle;
* Left Ventricle Ejection fraction < 10%;
* Unstable angina;
* Severe aortic stenosis
* Primary severe mitral insufficiency;
* New York Heart Association (NYHA) functional class IV;
* Previous cardiac surgery or scheduled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Time to Ventricular Tachycardia Recurrence | 12 months
  Compare the time to the first documented Ventricular Tachycardia episode between groups
Burden of Ventricular Tachycardia Recurrence | 12 months
  Compare the number of Ventricular Tachycardia episodes between groups in 12 months

SECONDARY OUTCOMES:
Ventricular Tachycardia Recurrence Following Sympathectomy Compared to Catheter Ablation. | 12 months
  Time to first VT episode after sympathectomy compared to Catheter ablation
Mortality and Transplant Rate | 12 months
  To compare between groups the number of patients who died or received a cardiac transplant at the end of the follow-up
Ventricular Ectopic Beats Density | 12 months
  To evaluate the density of ventricular premature beats in the 24-hour Holter in the follow-up, for each group.
Length of Hospital Stay | 12 months
  Compare the number of in-hospital days according to the type of intervention.
Rate of Complications Following Intervention | 12 months
  Compare the rate of clinical complications according to the type of intervention.
Impact on Left Ventricular Ejection Fraction | 12 months
  To evaluate the variations of the Left Ventricular Ejection Fraction in each group.
Autonomic Measures | 12 months
  To compare the RR variability measures in the 24h-Holter between groups

CONTACTS AND LOCATIONS:
Overall Officials: Paulo M Pego Fernandes, MD, PhD, Principal Investigator — Instituto do Coração Faculdade de Medicina da USP - (INCOR-FMUSP); Rodrigo M Kulchetscki, MD, Principal Investigator — Instituto do Coração Faculdade de Medicina da USP - (INCOR-FMUSP); Maurício I Scanavacca, MD, PhD, Study Director — Instituto do Coração Faculdade de Medicina da USP - (INCOR-FMUSP)
Locations (1):
- Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with other investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years
Access Criteria: Upon request.